CLINICAL TRIAL: NCT02133495
Title: Use of Non-Cadaveric Human Acellular Dermal Tissue (BellaDerm®) in Lower Eyelid Retraction Repair
Brief Title: An Outcomes Assessment of the Utility of Belladerm Acellular Dermal Allograft in Ocular Lower Lid Retraction Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SGM Physician Research Consortium (Network)
Collaborators: Musculoskeletal Transplant Foundation (Other)
Responsible Party: Principal Investigator, Kenneth Morgenstern, MD, Kenneth Morgenstern, MD, SGM Physician Research Consortium
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMBella1
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Lower Eyelid Retraction
Keywords: lower eyelid; retraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label (Experimental): Non Cadaveric human BellaDerm Acellular dermal tissue
  Interventions: Procedure: Non Cadaveric Human Acellular Dermal Tissue

INTERVENTIONS:
Procedure: Non Cadaveric Human Acellular Dermal Tissue
  Other Names: Bella Derm

SUMMARY:
The purpose of this study is to Evaluate the efficacy and longevity of a Human-derived, non-cadaveric, acellular dermal implant (BellaDerm) as a posterior spacer graft in the correction of lower eyelid retraction, taking into consideration issues associated with the use of acelular dermis such as contraction and potential regression of repairs.

DETAILED DESCRIPTION:
To Evaluate the efficacy and longevity of a Human-derived, non-cadaveric, acellular dermal implant (BellaDerm) as a posterior spacer graft in the correction of lower eyelid retraction, taking into consideration issues associated with the use of acelular dermis such as contraction and potential regression of repairs.

ELIGIBILITY:
Inclusion Criteria:

* Lower eyelid retraction, defined as inferior displacement of the lower eyelid margin with inferior scleral show, may be asymptomatic
* May have ocular irritation including foreign body sensation, burning, photophobia and tearing.
* May have aesthetically unsatisfactory eyelid appearance.

Exclusion Criteria:

* Have a condition that would be contraindicated to surgery

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Pre and Post operative margin reflex distance 2 MRD 2 | 1 year
  Pre and postoperative margin reflex distance 2 (MRD2) and inferior scleral show (ISS) was measured of each eyelid, and success was defined as a positive eyelid elevation and decrease in inferior scleral show. Long- term stability beyond 12 months was evaluated.

OTHER OUTCOMES:
Inferior scleral show | 1 year
  Pre and post operative margin reflex distance 2 (MRD2) and inferior scleral show (ISS) where measured for each eyelid elevation and decrease in inferior scleral show.

CONTACTS AND LOCATIONS:
Locations (1):
- Morgenstern Center for Orbital and Facial Plastic Surgery, Wayne, Pennsylvania, United States